CLINICAL TRIAL: NCT05216523
Title: "Review of Barotrauma in Admitted Covid-19 Cases - A Single Center Retrospective Study From March 2020 Till April 2021."
Brief Title: "Barotrauma in Admitted Covid-19 Cases - A Single Center Retrospective Study"
Acronym: BARCOV
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr Jyoti Burad, Senior specialist, Sultan Qaboos University
Other Study IDs: #2463
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Barotrauma; COVID-19
Keywords: Barotrauma; COVID-19; positive pressure ventilation; ferritin; steroids
MeSH Terms: conditions — Barotrauma; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Admitted Covid-19 cases who developed Barotrauma
- Controls: Admitted Covid-19 cases who did not develop Barotrauma, matched with Cases with respect to age and sex.

SUMMARY:
A retrospective study is planned to find out the incidence and association type of respiratory support with barotrauma in Covid-19 cases admitted in Sultan Qaboos University Hospital. As widely known, Covid-19 affects the respiratory system primarily and is the main cause of admission to hospital. Depending upon the severity, different levels of respiratory support are offered to the patients. Normally patients with viral/bacterial respiratory diseases have a low incidence of barotrauma. Since this disease is new and it has been observed that a significant number of covid-19 patients develop barotrauma, hence it is deemed worthwhile to investigate the matter.

All the patients admitted to the ward, high dependency unit, and intensive care unit will be scanned and those who developed barotrauma (pneumothorax, surgical emphysema, pneumo-pericardium, and pneumo-mediastinum) will be studied in detail and analyzed.

This review is expected to highlight the problem and etiology and we might be able to suggest a management strategy to deal with this problem.

DETAILED DESCRIPTION:
Introduction

Covid-19 is a recently emerged disease affecting the respiratory system primarily but later on, progresses to multisystem involvement. Most of the cases are mild and self-remitting. However, those who develop moderate to severe symptoms require admission. They receive different modalities of respiratory support as per the international guidelines.

The covid-19 typically starts with mild respiratory symptoms with fever, headache, and myalgia. Most of the cases remit after these by 10 days, but around 15% progress to more severe symptoms such as worsening of fever, respiratory symptoms leading to hypoxemia proceeding to complications further on. Correspondingly, the radiological findings peak by 2 weeks after symptom onset. By this point in time, the patients start requiring respiratory support and complications start to emerge as the time passes. Bacterial superinfections, interleukin surge, septic shock are commonly encountered. Recently, at our center rising episodes of barotrauma have been observed.

In the covid era because of huge numbers of admissions, the hospital, as well as ICU beds with respiratory and monitoring resources, are becoming significantly scarce. Hence prevention of complications can have a great impact on improving patient outcomes and utilizing hospital resources.

There can be few recognized mechanisms of barotrauma in Covid-19 cases. One of them is alveolar overdistension leading to rupture and barotrauma and the second is a decrease in the caliber of pulmonary vessels increasing pressure gradient causing air leak to the sheath. Positive pressure ventilation leads to an increase in intra-alveolar alveoli. Macklin phenomenon also describes the occurrence of a large pressure gradient between marginal alveoli and lung interstitium leading to barotrauma.

Barotrauma is treated by intercostal drain insertion, as well as conservative management by the reduction in airway pressures and increase in oxygen supplementation. Both these can lead to setbacks in a patient's recovery.

This research will identify the etiology of barotrauma and will highlight the preventive strategy to deal with it.

Aim of the Study:

This study aims to examine the incidence of barotrauma, its association with different management strategies so as to suggest modification of preventive and inciting factors. This may improve patient outcomes and conserve hospital resources.

Specific objectives:

1. To study the incidence of barotrauma in hospitalized Covid-19 cases.
2. To find the association of factors inciting barotrauma.
3. To formulate a management plan for the prevention of barotrauma in these cases.

Methodology and study design:

This retrospective study will be conducted in the Department of Anesthesia and ICU at Sultan Qaboos University hospital (SQUH) situated in Muscat, Oman. All admitted patients of Covid-19/SARS-2 between March 2020 to April 2021 will be scanned in the computerized system with the keywords: barotrauma, pneumothorax, surgical emphysema, pneumo-pericardium, and pneumo-mediastinum. A list of cases with these problems will be obtained and the cases will be studied in detail. Data will be obtained from SQUH "Track Care" hospital information system.

Study Population:

Inclusions:

● All admitted patients of Covid-19/SARS-2 between March 2020 to April 2021 t SQUH

Exclusions:

● Patients who develop barotrauma due to central line insertion or trauma prior to admission.

Data Collection and Analyses:

Demographic details, Day of barotrauma, comorbidities, type of respiratory support, other treatment modalities, and covid laboratory profile: ferritin, LDH, CRP, IL-6, fibrinogen, white cell count, and lymphocyte counts.

SPSS software (version 23) will be used to collect and analyze data. Obtaining the significance of association will be through using students' t-test, fisher's exact test, and Chi-square test. P-value < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All admitted adult patients with covid PCR positive result
* Those who developed barotrauma were labeled as "Cases" and those without barotrauma were "Controls".

Exclusion Criteria:

* Adult patients with covid PCR positive result who were discharged from Emergency department.
* Adult patients with covid PCR positive result who died or left against medical advice before admission to ward/ICU
* Adult patients with covid PCR positive result who were shifted to other hospitals and their follow up could not be completed.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2159 Covid-19 PCR-positive patients were identified in consecutive participant sampling at the University hospital during the study period. Out of these 63 patients were found to develop barotrauma. Matched controls were identified and a total of 322 cases was scanned. 61 patients were discharged from the emergency department after initial treatment, 1 patient left against medical advice and 2 patients died before they could be admitted to the ward and 7 were shifted to other hospitals, and their follow-up was lost, hence a total of 251 patients were finally studied. 63 patients were "Cases" and 188 were "Controls" in the ratio of 1:3 cases: controls.
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Barotrauma in admitted Covid-19 cases | 1-102 days
  Incidence of Barotrauma in admitted Covid-19 cases between March 2020 till April 2021

SECONDARY OUTCOMES:
Association of factors with Barotrauma in admitted Covid-19 cases | 1-102 days
  Association of factors with Barotrauma in admitted Covid-19 cases
Mortality with cases versus controls | 1-102 days
  Mortality with cases versus controls
Ventilation days of cases versus controls | 1-65 days
  Ventilation days

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, Study Director — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Undecided
IPD might be made available on individual request

REFERENCES:
- [Background] Pascarella G, Strumia A, Piliego C, Bruno F, Del Buono R, Costa F, Scarlata S, Agro FE. COVID-19 diagnosis and management: a comprehensive review. J Intern Med. 2020 Aug;288(2):192-206. doi: 10.1111/joim.13091. Epub 2020 May 13. PMID 32348588
- [Background] Kanne JP, Bai H, Bernheim A, Chung M, Haramati LB, Kallmes DF, Little BP, Rubin GD, Sverzellati N. COVID-19 Imaging: What We Know Now and What Remains Unknown. Radiology. 2021 Jun;299(3):E262-E279. doi: 10.1148/radiol.2021204522. Epub 2021 Feb 9. PMID 33560192
- [Background] Supady A, Curtis JR, Abrams D, Lorusso R, Bein T, Boldt J, Brown CE, Duerschmied D, Metaxa V, Brodie D. Allocating scarce intensive care resources during the COVID-19 pandemic: practical challenges to theoretical frameworks. Lancet Respir Med. 2021 Apr;9(4):430-434. doi: 10.1016/S2213-2600(20)30580-4. Epub 2021 Jan 12. PMID 33450202
- [Background] Elhakim TS, Abdul HS, Pelaez Romero C, Rodriguez-Fuentes Y. Spontaneous pneumomediastinum, pneumothorax and subcutaneous emphysema in COVID-19 pneumonia: a rare case and literature review. BMJ Case Rep. 2020 Dec 12;13(12):e239489. doi: 10.1136/bcr-2020-239489. PMID 33310838